CLINICAL TRIAL: NCT02371096
Title: Comparative Pharmacokinetic Trial of RGB-03 and MabThera
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gedeon Richter Plc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RGB-03-104
Record Dates: First submitted 2015-02-05; First posted 2015-02-25 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RGB-03 (Experimental)
  Interventions: Drug: RGB-03
- MabThera (rituximab) (Active Comparator)
  Interventions: Drug: MabThera (rituximab)

INTERVENTIONS:
Drug: MabThera (rituximab)
  Arms: MabThera (rituximab)
Drug: RGB-03
  Arms: RGB-03

SUMMARY:
Pharmacokinetic properties, efficacy, safety and tolerability of RGB-03 and MabThera will be compared in patients suffering from Rheumatoid Arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Active Rheumatoid Arthritis
* Inadequate response or intolerance to other DMARDs and anti-TNFs
* Treatment with Methotrexate

Exclusion Criteria:

* Previous treatment with rituximab
* Patients with systemic manifestations of rheumatoid arthritis
* Patients seropositive for HIV, HCV, HBV
* Female patients nursing

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Area under the serum concentration versus time curve (AUC) | 0-24 weeks